CLINICAL TRIAL: NCT02609399
Title: Influenza Therapeutic Trial: A Pilot Randomized Controlled Trial for Feasibility of Enrolling Subjects for Influenza Therapeutic Trials and Administering Influenza Antivirals in the Emergency Department to High Risk Subjects
Brief Title: ED Influenza Therapeutic Pilot Study: Oseltamivir vs. Peramivir
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: Department of Health and Human Services (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB00080405; 1 IDSEP150026-01-00 (Other Grant/Funding Number: Department of Health and Human Services); 1 IDSEP160031-01-00 (Other Grant/Funding Number: Department of Health and Human Services)
Record Dates: First submitted 2015-10-27; First posted 2015-11-20 (Estimated); Results first posted 2018-06-20 (Actual); Last update posted 2019-10-04 (Actual); Status verified 2019-09

CONDITIONS: Influenza
Keywords: Influenza; Antiviral treatment; Emergency department; Influenza therapeutics; Rapid influenza testing
MeSH Terms: conditions — Influenza, Human; Emergencies | interventions — Oseltamivir; peramivir

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Oseltamivir (Experimental): Subjects randomized to the oral treatment arm will receive 5 days of oral oseltamivir.
  Interventions: Drug: Oseltamivir
- Peramivir (Experimental): Subjects randomized to the IV treatment group will receive 1 dose of IV peramivir.
  Interventions: Drug: Peramivir

INTERVENTIONS:
Drug: Oseltamivir — Oral
  Other Names: Tamiflu
  Arms: Oseltamivir
Drug: Peramivir — IV
  Note: Subjects admitted to the hospital directly from the ED Enrollment Visit may receive more doses at the discretion of the treating physician.
  Other Names: Rapivab
  Arms: Peramivir

SUMMARY:
This pilot study is designed to demonstrate the feasibility of utilizing Emergency Departments (EDs) as a primary site for subject enrollment in clinical trials evaluating influenza therapeutics, and to provide pilot data for future clinical trial design and planning.

Primary Objective: To prospectively enroll high-risk subjects with laboratory-confirmed influenza into a randomized, open label study of oral versus IV influenza therapeutic to include symptom evaluation and outcome assessments.

Secondary Objective 1: To identify influenza positive patients utilizing a previously established triage-based assessment and rapid testing algorithm for suspected influenza infection.

Secondary Objective 2: To retrospectively evaluate all potentially eligible patients for potential enrollment biases.

Secondary Objective 3: To create a repository of residual nasopharyngeal samples collected from ED patients with suspected influenza illness.

DETAILED DESCRIPTION:
Title: A Pilot Randomized Controlled Trial for Feasibility of Enrolling Subjects for Influenza Therapeutic Trials and Administering Influenza Antivirals in the Emergency Department to High Risk Subjects

Population: Adults presenting to the emergency department (ED) with laboratory confirmed influenza who meet Centers for Disease Control and Prevention (CDC) criteria for antiviral treatment

Informed consent: Written informed consent

Number of Sites: 2 - large, urban, academically-affiliated, US EDs

Study Duration: November 2015 - June 2018

Subject Participation Duration: 4 weeks

Description of Agent or Intervention: Subjects will be randomized to either oral (oseltamivir) or intravenous (IV) (peramivir) antiviral treatment.

Description of Study Design: This is an open-label randomized controlled clinical trial in which subjects with influenza are randomized to either oral (oseltamivir) or IV (peramivir) antiviral treatment.

Estimated Time to Complete Enrollment: Subject enrollment will occur over two influenza seasons (November 2015 - April 2016 and November 2016 - April 2017) or longer, at the Principal Investigator's discretion, based on influenza prevalence.

ELIGIBILITY:
Inclusion Criteria:

* Eligible patients include all patients who present to the emergency department (ED) between November and April of each influenza season, or later, at the Co-PIs' discretion, based on influenza prevalence, with the following criteria:

  1. 18 years of age or older
  2. Laboratory confirmed positive influenza test associated with their current ED visit
  3. Symptoms of acute respiratory illness for ≤4 days (96 hours)
  4. Meets CDC criteria for antiviral treatment
* For the purpose of this study, acute respiratory illness is defined as presence of any of the following symptoms: new or increased cough, new or increased shortness of breath, change in sputum production (for adults 65 years or older), sinus pain, nasal congestion, rhinorrhea, sore throat, subjective fever reported at time of triage or documented fever (defined here as ≥ 38 degrees Celsius).
* CDC criteria for influenza antiviral treatment is defined as: being age 65 years old or older, pregnant or less than two weeks postpartum, American Indian or Alaska native, morbid obesity (BMI ≥40), a current resident of nursing home or other chronic-care facility, having chronic pulmonary disease, cardiovascular disease (except hypertension alone), renal disease, hepatic disease, hematologic disease, metabolic disorders, neurologic and neurodevelopment conditions, immunosuppression (including that caused by medications or by HIV infection), being admitted to inpatient or an observation unit, or having a clinical diagnosis of pneumonia (by the ED physician).

Exclusion Criteria:

1. Does not speak and understand English (or English or Spanish)
2. Unable or unwilling to provide informed consent
3. Previously enrolled in the study during the current influenza season
4. Unable to take oral medication
5. Unable to comply with all planned study procedures including availability for follow-up and willingness to complete study diary and self-assessment
6. Use of neuraminidase inhibitors within the past seven days
7. Known allergic reaction to neuraminidase inhibitors
8. Pregnant or breastfeeding
9. End-stage renal disease, defined as 9a. Currently undergoing dialysis (either hemo or peritoneal); or 9b. Creatinine clearance (CrCl) of <10 mL/min.
10. End-stage liver disease, as determined by the treating ED provider
11. Glucose-6-phosphate dehydrogenase (G6PD) deficiency by patient report
12. Immunodeficiency, defined as:

12a. Solid organ transplant patients receiving immunosuppression; 12b. Hematopoietic stem cell transplant patients within 12 months of transplant or with ongoing immunosuppression; 12c. Oncology patients who have had chemotherapy within the past 30 days; 12d. Current treatment with steroids equivalent to 10 mg of prednisone or more per day for greater than two weeks; 12e. Rheumatologic patients receiving immunosuppressive therapy; or 12f. HIV patients who meet one of the following criteria: 12fi. Have a cluster of differentiation 4 (CD4) cell count of <200 cells/mm3 within the past 3 months ; 12fii. Not actively receiving highly active antiretroviral therapy (HAART); or 12fiii. Have an absolute lymphocyte count <1.0 x 103 cells/μL conducted at the current ED visit

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Actual)
Dates: Start 2015-11-01 (Actual); Primary Completion 2017-05-26 (Actual); Study Completion 2018-05-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Richard Rothman, MD, PhD, Principal Investigator — Johns Hopkins University
Locations (2):
- United States (2):
  - Maricopa Integrated Health System, Phoenix, Arizona
  - Johns Hopkins Hospital, Baltimore, Maryland

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study recruited adult patients through both clinical testing and screening with a Clinical Decision Guideline (CDG) over two influenza seasons at the following academically affiliated U.S. Emergency Departments (EDs):
  * November 2015- April 2016: Johns Hopkins Hospital (JHH)
  * November 2016- April 2017: JHH and Maricopa Medical Center (MMC)
Groups:
- Peramivir: Subjects randomized to the IV treatment group will receive 1 dose of IV peramivir. (Subjects admitted to the hospital directly from the ED Enrollment Visit may receive more doses at the discretion of the treating physician).
Period: Influenza Season 2015-2016
Arm/Group | Oseltamivir | Peramivir
Started | 27 | 31
Completed | 24 | 29
Not Completed | 3 | 2
Not completed — Lost to Follow-up | 3 | 2
Period: Influenza Season 2016-2017
Arm/Group | Oseltamivir | Peramivir
Started | 58 | 64
Completed | 49 | 59
Not Completed | 9 | 5
Not completed — Lost to Follow-up | 8 | 5
Not completed — Found ineligible after randomization | 1 | 0

BASELINE CHARACTERISTICS:
Population: For baseline analyses, overall characteristics (seasons 2015-2016 & 2016-2017) & characteristics stratified by influenza season (2015-2016 vs. 2016-2017) are presented. Total number of subjects contributing data to 2015-2016 baseline analyses was 58, compared to 121 subjects for 2016-2017 season. Information unavailable: 1 oseltamivir participant
Groups:
- Experimental: Oseltamivir: Subjects randomized to the oral treatment arm will receive 5 days of oral oseltamivir.
- Experimental: Peramivir: Subjects randomized to the IV treatment group will receive 1 dose of IV peramivir.
- Total: Total of all reporting groups
Arm/Group | Experimental: Oseltamivir | Experimental: Peramivir | Total
Number analyzed (Participants) | 84 | 95 | 179
Age, Continuous [Mean (Full Range); unit: years] — Baseline measures includes both influenza seasons 2015-2016 and 2016-2017. A total of 180 subjects were enrolled across both seasons. Baseline information is unavailable for 1 participant in the oseltamivir arm
  years | 47.3 [20 to 78] | 47.5 [19 to 80] | 47.4 [19 to 80]
Sex: Female, Male [Count of Participants; unit: Participants] — Baseline measures includes both influenza seasons 2015-2016 and 2016-2017. A total of 180 subjects were enrolled across both seasons. Baseline information is unavailable for 1 participant in the oseltamivir arm
  Participants
    Female | 48 | 58 | 106
    Male | 36 | 37 | 73
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Baseline measures includes both influenza seasons 2015-2016 and 2016-2017. A total of 180 subjects were enrolled across both seasons. Baseline information is unavailable for 1 participant in the oseltamivir arm
  Participants
    Hispanic or Latino | 10 | 19 | 29
    Not Hispanic or Latino | 74 | 76 | 150
    Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants] — Baseline measures includes both influenza seasons 2015-2016 and 2016-2017. A total of 180 subjects were enrolled across both seasons. Baseline information is unavailable for 1 participant in the oseltamivir arm
  Participants
    American Indian or Alaska Native | 1 | 2 | 3
    Asian | 2 | 1 | 3
    Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
    Black or African American | 60 | 60 | 120
    White | 21 | 29 | 50
    More than one race | 0 | 0 | 0
    Unknown or Not Reported | 0 | 3 | 3
Region of Enrollment [Number; unit: participants]
  United States | 84 | 95 | 179
Age, Continuous (Influenza Season 2015-2016) [Mean (Full Range); unit: years] — Population: This measure is specific to the 2015-2016 influenza season, during which 58 subjects were enrolled and analyzed.
  years
    number analyzed (Participants) | 27 | 31 | 58
    (all) | 48.7 [20 to 68] | 43.7 [19 to 72] | 46 [19 to 72]
Age, Continuous (Influenza Season 2016-2017) [Mean (Full Range); unit: years] — Population: This measure is specific to the 2016-2017 influenza season, during which 122 subjects were enrolled and analyzed. Baseline information is unavailable for 1 participant in the oseltamivir arm.
  years
    number analyzed (Participants) | 57 | 64 | 121
    (all) | 46.6 [20 to 78] | 49.3 [20 to 80] | 48.0 [20 to 80]
Sex: Female, Male (Influenza Season 2015-2016) [Count of Participants; unit: Participants] — Population: This measure is specific to the 2015-2016 influenza season, during which 58 subjects were enrolled and analyzed.
  Participants
    number analyzed (Participants) | 27 | 31 | 58
    Female | 11 | 17 | 28
    Male | 16 | 14 | 30
Sex: Female, Male (Influenza Season 2016-2017) [Count of Participants; unit: Participants] — Population: This measure is specific to the 2016-2017 influenza season, during which 122 subjects were enrolled and analyzed. Baseline information is unavailable for 1 participant in the oseltamivir arm
  Participants
    number analyzed (Participants) | 57 | 64 | 121
    Female | 37 | 41 | 78
    Male | 20 | 23 | 43
Ethnicity (NIH/OMB) (Influenza Season 2015-2016) [Count of Participants; unit: Participants] — Population: This measure is specific to the 2015-2016 influenza season, during which 58 subjects were enrolled and analyzed.
  Participants
    number analyzed (Participants) | 27 | 31 | 58
    Hispanic or Latino | 0 | 0 | 0
    Not Hispanic or Latino | 27 | 31 | 58
Ethnicity (NIH/OMB) (Influenza Season 2016-2017) [Count of Participants; unit: Participants] — Population: This measure is specific to the 2016-2017 influenza season, during which 122 subjects were enrolled and analyzed. Baseline information is unavailable for 1 participant in the oseltamivir arm
  Participants
    number analyzed (Participants) | 57 | 64 | 121
    Hispanic or Latino | 10 | 19 | 29
    Not Hispanic or Latino | 47 | 45 | 92
Race (NIH/OMB) (Influenza Season 2015-2016) [Count of Participants; unit: Participants] — Population: This measure is specific to the 2015-2016 influenza season, during which 58 subjects were enrolled and analyzed.
  Participants
    number analyzed (Participants) | 27 | 31 | 58
    American Indian or Alaska Native | 0 | 1 | 1
    Asian | 0 | 1 | 1
    Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
    Black or African American | 22 | 24 | 46
    White | 5 | 5 | 10
    More than one race | 0 | 0 | 0
    Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) (Influenza Season 2016-2017) [Count of Participants; unit: Participants] — Population: This measure is specific to the 2016-2017 influenza season, during which 122 subjects were enrolled and analyzed. Baseline information is unavailable for 1 participant in the oseltamivir arm
  Participants
    number analyzed (Participants) | 57 | 64 | 121
    American Indian or Alaska Native | 1 | 1 | 2
    Asian | 2 | 0 | 2
    Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
    Black or African American | 38 | 36 | 74
    White | 16 | 24 | 40
    More than one race | 0 | 0 | 0
    Unknown or Not Reported | 0 | 3 | 3

OUTCOME MEASURES:

1. Primary Outcome: Mean Symptom Severity Score During the 2015-2016 Influenza Season for Symptom Domains as Assessed Using the Influenza-Patient Reported Outcome (FLU-PRO™) Questionnaire
Description: Symptom evaluation during the 2015-2016 influenza season as recorded through FLU-PRO™: a daily diary developed to assess occurrence and severity of influenza symptoms.
  Item responses:
  1. Not at all
  2. A little bit
  3. Somewhat
  4. Quite a bit
  5. Very much
Time Frame: ED Enrollment Visit through Day 14 ( 2015-2016 influenza season)
Population: All subjects enrolled and randomized.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Oseltamivir | Peramivir
Number analyzed (Participants) | 27 | 31
units on a scale
  Nose | 1.4 (0.8) | 1.9 (1.3)
  Throat | 1.3 (0.8) | 1.7 (1.2)
  Eyes | 1.2 (0.6) | 1.6 (1.2)
  Chest/Respiratory | 1.9 (1.2) | 2.3 (1.5)
  Gastrointestinal | 1.5 (1.1) | 1.5 (1.1)
  Body/Systemic | 1.7 (1.2) | 1.9 (1.4)
  Total/Overall | 1.6 (1.1) | 1.9 (1.4)

2. Primary Outcome: Mean Symptom Severity Score During the 2016-2017 Influenza Season for Symptom Domains as Assessed Using the FLU-PRO™ Questionnaire
Description: Symptom evaluation during the 2016-2017 influenza season as recorded through FLU-PRO™: a daily diary developed to assess occurrence and severity of influenza symptoms.
  Item responses:
  1. Not at all
  2. A little bit
  3. Somewhat
  4. Quite a bit
  5. Very much
Time Frame: ED Enrollment Visit through Day 14 ( 2016-2017 influenza season)
Population: All enrolled and randomized subjects with the exception of 1 inadvertent enrollment (subject found to be ineligible shortly after randomization)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Oseltamivir | Peramivir
Number analyzed (Participants) | 57 | 64
units on a scale
  Nose | 1.5 (0.8) | 1.5 (0.7)
  Throat | 1.3 (0.6) | 1.4 (0.8)
  Eyes | 1.3 (0.7) | 1.2 (0.5)
  Chest/Respiratory | 1.7 (0.8) | 1.8 (0.9)
  Gastrointestinal | 1.3 (0.7) | 1.3 (0.7)
  Body/Systemic | 1.5 (0.8) | 1.5 (0.8)
  Total/Overall | 1.4 (0.6) | 1.5 (0.6)

3. Primary Outcome: Mean Karnofsky Performance Scale Score During the 2015-2016 Influenza Season
Description: The Karnofsky Performance Scale is a tool for assessing subject functional impairment.
  Subjects provided or received (from a healthcare provider such as a doctor or nurse) a daily rating from 0 (Dead) to 100 (Normal - no complaints, no evidence of disease) from enrollment through Day 14 of the 2015-2016 influenza season.
Time Frame: ED Enrollment Visit through Day 14 ( 2015-2016 influenza season)
Population: All subjects enrolled and randomized.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Experimental: Oseltamivir: Subjects randomized to the oral treatment arm received 5 days of oral oseltamivir.
- Experimental: Peramivir: Subjects randomized to the IV treatment group will receive 1 dose of IV peramivir. (Subjects admitted to the hospital directly from the ED Enrollment Visit may receive more doses at the discretion of the treating physician).
Arm/Group | Experimental: Oseltamivir | Experimental: Peramivir
Number analyzed (Participants) | 27 | 31
units on a scale | 77.1 (20.8) | 73.2 (19.9)

4. Primary Outcome: Mean Karnofsky Performance Scale Score During the 2016-2017 Influenza Season
Description: The Karnofsky Performance Scale is a tool for assessing subject functional impairment.
  Subjects provided or received (from a healthcare provider such as a doctor or nurse) a daily rating from 0 (Dead) to 100 (Normal - no complaints, no evidence of disease) from enrollment through Day 14 of the 2016-2017 influenza season.
Time Frame: ED Enrollment Visit through Day 14 ( 2016-2017 influenza season)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Experimental: Oseltamivir | Experimental: Peramivir
Number analyzed (Participants) | 57 | 64
units on a scale | 80.0 (10.7) | 79.9 (9.1)

ADVERSE EVENTS:
Time Frame: Accrual for the 2015-2016 influenza season opened on 11/1/2015 and closed on 4/30/2016. Accrual for the 2016-2017 influenza season opened on 11/1/2016 and closed on 4/30/2017. All enrolled participants were assessed for adverse events from enrollment visit until the end of study follow up on Day 28.
Groups:
- Peramivir: Subjects randomized to the IV treatment group will receive 1 dose (or more as appropriate at the discretion of the treating physician) of IV peramivir.
  Peramivir: IV
  Note: Should a patient remain in the hospital after 5 days of treatment, and the patient is symptomatically better, treatment will stop. If the patient remains hospitalized after 5 days of treatment and has not improved, the treating physician will continue to have an option to continue use of peramivir daily for another 5 day course.
Arm/Group | Oseltamivir | Peramivir
All-Cause Mortality (participants affected / at risk) | 0/84 | 0/95
Serious Adverse Events (participants affected / at risk) | 4/84 | 9/95
Other Adverse Events (participants affected / at risk) | 49/84 | 54/95
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Oseltamivir (N=84) | Peramivir (N=95)
Intestinal perforation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Blood creatinine increased (Investigations) | 1 (1) | 0 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Myocardial infarction (Cardiac disorders) | 0 (0) | 1 (1)
Coronary artery disease (Cardiac disorders) | 0 (0) | 1 (1)
Hypotension (Vascular disorders) | 0 (0) | 2 (2)
Syncope (Nervous system disorders) | 0 (0) | 1 (1)
Facial paralysis (Nervous system disorders) | 0 (0) | 1 (1)
Abdominal Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Chronic obstructive pulmonary disease (COPD) (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pre-op admission (Surgical and medical procedures) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Oseltamivir (N=84) | Peramivir (N=95)
Diarrhea (Gastrointestinal disorders) | 28 (32) | 31 (36)
Nausea (Gastrointestinal disorders) | 27 (29) | 21 (23)
Vomiting (Gastrointestinal disorders) | 19 (20) | 16 (17)
Insomnia (Psychiatric disorders) | 12 (14) | 18 (18)
Rash (Skin and subcutaneous tissue disorders) | 7 (8) | 5 (6)
Vertigo (Ear and labyrinth disorders) | 9 (9) | 10 (12)
Confusion/Hallucinations (Nervous system disorders) | 6 (6) | 7 (7)

LIMITATIONS AND CAVEATS:
1. Not designed or powered to assess differences in clinical outcomes.
2. Planned to recruit >= 50 subjects/site, but MMC enrolled 44 due to lower-than-expected flu incidence and Hopkins Uni. increased enrollment to make up for the shortfall.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2016-09-26): https://cdn.clinicaltrials.gov/large-docs/99/NCT02609399/Prot_SAP_ICF_003.pdf